CLINICAL TRIAL: NCT01703936
Title: Evaluating a Landmine Action Ex-combatant Reintegration Program in Liberia
Brief Title: Ex-combatant Reintegration in Liberia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: United Nations (Other); World Bank (Other)
Responsible Party: Principal Investigator, Christopher J. Blattman, Assistant Professor of International and Public Affairs and of Political Science, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: AAAK6203
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Poverty; Social Instability
Keywords: economic intervention; ex-combatant; agriculture; life skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- agricultural training program (Experimental): Three to four month residential agriculture and life skills training program.
  Interventions: Other: Agricultural and life skills training program
- Control group (No Intervention)

INTERVENTIONS:
Other: Agricultural and life skills training program
  Other Names: Tumutu Agricultural Training Program (TATP); Sinoe Agricultural Training Program (SATP)
  Arms: agricultural training program

SUMMARY:
This project is an evaluation of an agricultural training and resettlement program for high-risk young adults in Liberia, especially poorly integrated male ex-combatants. The primary aim is to see to what extent an intensive economic and life skills intervention can rehabilitate high-risk individuals and reduce aggression and armed violence.

DETAILED DESCRIPTION:
Poor and unemployed youth are widely considered a threat to political stability, often blamed for everything from fights to crime, riots and revolutions. Ex-combatants cause special worry. Not only do they have professional experience in warfare, and hence some comparative advantage in violence, but their social networks may also be dense with potential recruiters. War may also have left them poorer or more traumatized than their peers. Each of these factors could elevate the risk of rebellion, crime, or other aggression, risks greatest in weak states and uncertain economic climates like that of Liberia.

In response, policymakers commonly turn to employment and other poverty alleviation programs, including cash grants, vocational training, small business development, and microfinance. Underlying these programs is the belief that with economic opportunities come stability. When dealing with organized populations, such as former combatants, gang members, or criminal organizations, policymakers are also anxious to break down risky social networks, especially the links between commanders and foot soldiers. Interventions often go beyond simple employment programs, and seek to relocate, resettle, or otherwise remove high-risk individuals from risky networks.

This project evaluates a rehabilitation program for ex-combatants and other high-risk youth in Liberia, a unique case where it was both politically and practically feasible to establish and follow a random control group. The program we study, which was designed and implemented by the international non-governmental organization (NGO) Action on Armed Violence, is among the best of its class. The program is targeted towards ex-combatants and other high-risk populations in resource enclaves and other "hotspots" around the country. It provides extensive agricultural skills training and inputs alongside life skills training and resettlement assistance. Its objective is to reduce the risk of violence and aggression by providing an alternative, stable livelihood in civilian communities to youth otherwise engaged in illicit activities or thought to be easily mobilized into crime or violence. After observing two highly promising courses and classes of graduates, the researchers collaborated with the NGO to randomly evaluate their next round of classes at two training sites.

The program implementers confirmed that the number of youth eligible for the program exceeded program capacity by a factor of at least two. The sample size was limited to 2.5 times the number of spots in the program, for a total of 1500. In order to give all eligible youth an equal opportunity to participate, the program implementers determined entry into the program using a computerized randomization of eligible youth. Respondents were assigned to treatment and control using a randomization program coded in Stata. The sample was stratified by gender, "commander status," and community of registration.

The study has two principal rounds of data collection among both treatment and control groups: a baseline prior to the intervention and a follow-up survey approximately one year following completion of the program.

ELIGIBILITY:
Inclusion Criteria (determined by program):

* ex-combatant
* not served by previous reintegration programs
* engaged in illicit activities such as mining and rubber tapping

Exclusion Criteria (determined by program):

* pregnant women
* individuals deemed physically incapable of agriculture
* foreigners unwilling to settle in Liberia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1330 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Potential for Social Instability | 1 year after completion of program
  This outcome includes engagement in illicit activities, ease of mobilization, political attitudes, violence and aggression, how settled they are, integration into mainstream society, and mental health symptoms.
Economic Stability | 1 year after completion of program
  This outcome includes employment and poverty level.
Preferences | 1 year after completion of program
  This outcome includes risk and time preferences.
Interest in Agriculture | 1 year after completion of the program
  This outcome measures level of interest in agriculture, attempts to engage in agriculture, perceptions of agriculture, and level of willingness to invest in agriculture.

SECONDARY OUTCOMES:
Level of Social Support and Quality of Social Relations | 1 year after completion of the study
  The outcome includes aggregate level of social support, quality of relationship with family and elders, advising, and peer groups.
Aspirations and Future Planning | 1 year after completion of the program
  This outcome measures aspirations for the future and thinking about the future.
Empowerment | 1 year after completion of the study
  The outcome includes locus of control and making their own decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie Annan, Ph.D., Principal Investigator — International Rescue Committee; Christopher Blattman, Ph.D., Principal Investigator — Columbia University
Locations (2):
- Liberia (2):
  - Tumutu Agricultural Training Program, Salala, Bong County
  - Sinoe Agricultural Training Program, Panama, Sinoe County

REFERENCES:
- See also: Related Info — http://poverty-action.org/project/0138